CLINICAL TRIAL: NCT03301701
Title: Randomized Feasibility Trial of Prostate Radiotherapy vs Prostatectomy in Men With Hormone Sensitive Oligometastatic Prostate Cancer
Brief Title: Feasibility Trial in Men With Hormone Sensitive Oligometastatic Prostate Cancer
Acronym: PRORAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accruals
Sponsor: Dr. Patrick Cheung (Other)
Responsible Party: Sponsor-Investigator, Dr. Patrick Cheung, Dr. Patrick Cheung, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRORAD
Record Dates: First submitted 2017-01-11; First posted 2017-10-04 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Hormone Sensitive Oligometastatic Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Radical prostatectomy
  Interventions: Procedure: Radical prostatectomy
- Arm 2 (Active Comparator): Radiotherapy
  Interventions: Radiation: HDR (19Gy) or SBRT (35-40Gy)

INTERVENTIONS:
Procedure: Radical prostatectomy — Radical prostatectomy
  Arms: Arm 1
Radiation: HDR (19Gy) or SBRT (35-40Gy) — Patients will receive HDR unless judged to medically unfit to undergo HDR brachytherapy, in which case they will receive SBRT
  Arms: Arm 2

SUMMARY:
Patients with hormone sensitive oligometastatic prostate cancer (≤ 5 metastatic tumours outside of regional pelvic nodes with no more than 3 in any organ system) and no previous treatment to prostate will be treated with intermittent androgen deprivation therapy +/- chemotherapy, stereotactic radiotherapy to all metastases, and either radical prostatectomy or radiotherapy.

DETAILED DESCRIPTION:
Investigators propose to do a randomized feasibility trial comparing RP vs RT to the prostate in the setting of hormone sensitive oligometastatic prostate cancer. SBRT will be used to treat all of the metastases, and this will be combined with an intermittent ADT approach. Adding systemic chemotherapy will be allowed. Given the past difficulties of randomizing patients between RP and RT in localized prostate cancer studies (like SPIRIT), investigators feel a small feasibility project is the first step. In the setting of metastatic disease, where radical treatment is not routine standard of care, we hope that patients will be more inclined to accept randomization. If patients do not accept their assigned randomization (ie they prefer RP even though they are randomized to RT, or vice versa), they will still be treated with their prostate intervention of choice and followed for their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Histologic confirmation of prostate adenocarcinoma.
* Stage IV disease with ≤ 5 metastases outside of the pelvis.
* ≤ 3 metastases in any one organ system.
* ECOG performance 0-1.
* All metastatic tumours amenable to SBRT.
* Patient eligible for either RP or RT to the prostate.

Exclusion Criteria:

* Castration resistant prostate cancer.
* Previous RP or RT to prostate.
* Inability to treat all metastases with SBRT.
* Prior malignancy within the past 5 years, excluding non-melanoma skin cancer, in-situ cancer, superficial bladder cancer, chronic lymphocytic leukemia or low grade lymphoma which is being observed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Patients willing to accept their randomization | 2 years
  Patients willing to accept their randomization will be measured as a proportion.

SECONDARY OUTCOMES:
Toxicity | 7 years
  Acute and late toxicities will be measured using CTCAE v4.0 and will be reported as percentages.
Efficacy | 7 years
  Time to CRPC will be calculated using Kaplan Meier methodology.
Efficacy | 7 years
  Progression free survival will be calculated using Kaplan Meier methodology.
Efficacy | 7 years
  Local control will be calculated using Kaplan Meier methodology.
Efficacy | 7 years
  Distant control will be calculated using Kaplan Meier methodology.
Efficacy | 7 years
  Overall survival will be calculated using Kaplan Meier methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cheung, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No